CLINICAL TRIAL: NCT06228586
Title: A Phase III, Open-label, Single-center Study to Describe the Immunogenicity and Safety of a Single Dose of MenACYW Conjugate Vaccine in Participants Aged 12 Months and Older in Vietnam
Brief Title: Study on a MenACYW Conjugate Vaccine Administered as a Single Dose in Participants Aged 12 Months and Older in Vietnam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEQ00074; U1111-1256-9172 (Registry Identifier: ICTRP); 2021-001699-41 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Meningococcal Infection; Healthy Volunteers
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MenACYW conjugate vaccine (Experimental): MenACYW conjugate vaccine single injection on Day 01
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine — Pharmaceutical form:Liquid solution-Route of administration:Intramuscular injection
  Other Names: MenACYW conjugate vaccine, MenQuadfi™

SUMMARY:
The MEQ00074 study was a Phase III, open-label, single-center study aimed at describing the immunogenicity and safety of a single dose of investigational quadrivalent Meningococcal Polysaccharide (serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine (MenACYW conjugate vaccine) in participants aged 12 months and older in Vietnam.

The primary objectives of the study were:

* To describe the antibody responses to meningococcal serogroups A, C, W, and Y before and 30 days after the administration of a single dose of MenACYW conjugate vaccine
* To describe the safety profile of a single dose of MenACYW conjugate vaccine The duration of each participant's participation will be approximately 30 to 44 days.

DETAILED DESCRIPTION:
The duration of each participant's participation was approximately 30 to 44 days.

ELIGIBILITY:
Inclusion Criteria:

- Aged 12 months and above on the day of inclusion

Adults:

* Aged 18 and above on the day of inclusion
* A female participant was eligible to participate if she was not pregnant or breastfeeding and one of the following conditions applies:

  * Was of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.
  * OR Was of childbearing potential and agreed to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential would have a negative highly sensitive pregnancy test (urine) within 1 week before the dose of study intervention.

* Informed consent form was signed and dated
* Was able to attend all scheduled visits and to comply with all study procedures

Adolescents:

* Aged 10 to 17 years on the day of inclusion
* A female participant was eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Was of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarche.
  * OR Was of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential would have a negative highly sensitive pregnancy test (urine) within 1 week before the dose of study intervention.

* Informed consent form was signed and dated by both the participant and the parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations Assent form was signed and dated by the participant (assent form required for participants aged 12 to 15 years) or verbal consent was obtained (for participants aged 10 to 11 years), and informed consent form was signed and dated by the parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and to comply with all study procedures

Children:

* Aged 2 to 9 years on the day of inclusion
* Verbal consent was obtained (for participants aged 7 to 9 years), and informed consent form was signed and dated by the parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and to comply with all study procedures

Toddlers

* Aged 12 to 23 months on the day of inclusion
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative and by an independent witness if required by local regulations
* Participant and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria apply:

Adults (aged 18 years and above), Adolescents (aged 10 to 17 years), Children (aged 2 to 9 years) and Toddlers (aged 12 to 23 months)

* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 4 weeks following study intervention administration except for influenza vaccination, which may be received at least 2 weeks before or after study vaccine. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (ie, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, W, or Y; or meningococcal B serogroup-containing vaccine)
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* History of any N. meningitidis infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal disease during the study (specifically but not limited to participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease)
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Personal history of Guillain-Barré syndrome (GBS)
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.5 C) or hypothermia (axillary temperature ≤ 35.5 C) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw

Adults (aged 18 years and above) and Adolescents (aged 10 to 17 years)

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoidcontaining vaccine within at least 10 years of the proposed study vaccination
* Self-reported thrombocytopenia, contraindicating intramuscular injection
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Children (aged 2 to 9 years)

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine
* Thrombocytopenia as reported by the parent/legally acceptable representative, or suspected thrombocytopenia contraindicating intramuscular injection
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

Toddlers (aged 12 to 23 months)

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine
* Thrombocytopenia as reported by the parent/legally acceptable representative, or suspected thrombocytopenia contraindicating intramuscular injection
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Vietnam (4):
  - Investigational Site Number : 7040001, Hanoi
  - Investigational Site Number : 7040002, Thái Bình
  - Investigational Site Number : 7040003, Thái Bình
  - Investigational Site Number : 7040004, Thái Bình

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: MEQ00074 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25592&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 investigational sites (1 main site and 3 satellite sites) in Vietnam from 18 January 2024 to 31 March 2024.
Pre-assignment Details: A total of 447 participants (223 participants aged 12-23 months and 224 participants aged >=24 months) were enrolled in this study.
Groups:
- MenACYW Conjugate Vaccine: 12-23 Months of Age: Participants aged 12-23 months received a single dose of 0.5 milliliter (mL) meningococcal polysaccharide (serogroups A, C, W, and Y) tetanus toxoid conjugate vaccine (MenACYW conjugate vaccine) as an intramuscular (IM) injection on Day 1.
- MenACYW Conjugate Vaccine: 24 Months of Age and Above: Participants aged >=24 months received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 1.
Period: Overall Study
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Started | 223 | 224
Vaccinated | 223 | 223
Completed | 220 | 223
Not Completed | 3 | 1
Not completed — Withdrawal by Participant or Parent/Guardian | 3 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled study participants were participants that had their eligibility evaluation and passed screening.
Groups:
- MenACYW Conjugate Vaccine: 12-23 Months of Age: Participants aged 12-23 months received a single dose of 0.5 mL MenACYW conjugate vaccine as an IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above | Total
Number analyzed (Participants) | 223 | 224 | 447
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 223 | 121 | 344
  Between 18 and 65 years | 0 | 88 | 88
  >=65 years | 0 | 15 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 130 | 248
  Male | 105 | 94 | 199
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W was measured in a serum bactericidal assay utilizing the human complement (hSBA).
Time Frame: Day 1 (pre-vaccination) and Day 31 (30 days post-vaccination on Day 1)
Population: Analysis was performed on the per-protocol analysis set (PPAS) which was a subset of the full analysis set (FAS). The FAS included participants who received the study vaccine and had a valid post-vaccination serology result.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 200 | 221
titer
  Serogroup A: Day 1 | 4.44 [4.00 to 4.92] | 7.58 [6.76 to 8.51]
  Serogroup A: Day 31 | 39.0 [32.9 to 46.2] | 43.2 [34.6 to 54.1]
  Serogroup C: Day 1 | 2.61 [2.34 to 2.91] | 5.65 [4.82 to 6.62]
  Serogroup C: Day 31 | 1226 [1076 to 1398] | 895 [781 to 1026]
  Serogroup Y: Day 1 | 2.86 [2.55 to 3.20] | 4.08 [3.47 to 4.78]
  Serogroup Y: Day 31 | 132 [112 to 156] | 288 [244 to 340]
  Serogroup W: Day 1 | 2.26 [2.09 to 2.44] | 4.33 [3.81 to 4.92]
  Serogroup W: Day 31 | 99.4 [85.6 to 115] | 166 [139 to 198]

2. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement Titers >=4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W was measured by hSBA. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 1 (pre-vaccination) and Day 31 (30 days post-vaccination on Day 1)
Population: Analysis was performed on the PPAS which was a subset of the FAS. The FAS included participants who received the study vaccine and had a valid post-vaccination serology result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 200 | 221
percentage of participants
  Serogroup A | 81.5 [75.4 to 86.6] | 66.5 [59.9 to 72.7]
  Serogroup C | 99.5 [97.2 to 100] | 97.7 [94.8 to 99.3]
  Serogroup Y | 96.5 [92.9 to 98.6] | 95.5 [91.8 to 97.8]
  Serogroup W | 94.5 [90.4 to 97.2] | 95.5 [91.8 to 97.8]

3. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement Titers >=1:4 and >=1:8
Description: as for outcome 2
Time Frame: Day 1 (pre-vaccination) and Day 31 (30 days post-vaccination on Day 1)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 200 | 221
percentage of participants
  Serogroup A: Day 1: >=1:4 | 79.5 [73.2 to 84.9] | 94.1 [90.2 to 96.8]
  Serogroup A: Day 1: >=1:8 | 25.0 [19.2 to 31.6] | 59.7 [52.9 to 66.3]
  Serogroup A: Day 31: >=1:4 | 97.5 [94.3 to 99.2] | 89.1 [84.3 to 92.9]
  Serogroup A: Day 31: >=1:8 | 93.5 [89.1 to 96.5] | 84.6 [79.2 to 89.1]
  Serogroup C: Day 1: >=1:4 | 16.5 [11.6 to 22.4] | 64.3 [57.6 to 70.6]
  Serogroup C: Day 1: >=1:8 | 8.5 [5.0 to 13.3] | 38.5 [32.0 to 45.2]
  Serogroup C: Day 31: >=1:4 | 100 [98.2 to 100] | 100 [98.3 to 100]
  Serogroup C: Day 31: >=1:8 | 100 [98.2 to 100] | 100 [98.3 to 100]
  Serogroup Y: Day 1: >=1:4 | 21.0 [15.6 to 27.3] | 35.3 [29.0 to 42.0]
  Serogroup Y: Day 1: >=1:8 | 15.5 [10.8 to 21.3] | 26.2 [20.6 to 32.6]
  Serogroup Y: Day 31: >=1:4 | 99.5 [97.2 to 100] | 99.1 [96.8 to 99.9]
  Serogroup Y: Day 31: >=1:8 | 98.5 [95.7 to 99.7] | 99.1 [96.8 to 99.9]
  Serogroup W: Day 1: >=1:4 | 7.0 [3.9 to 11.5] | 51.6 [44.8 to 58.3]
  Serogroup W: Day 1: >=1:8 | 4.0 [1.7 to 7.7] | 32.1 [26.0 to 38.7]
  Serogroup W: Day 31: >=1:4 | 99.5 [97.2 to 100] | 100 [98.3 to 100]
  Serogroup W: Day 31: >=1:8 | 98.5 [95.7 to 99.7] | 100 [98.3 to 100]

4. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement Vaccine Seroresponse for Serogroups A, C, Y, and W
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W was measured by hSBA. hSBA vaccine seroresponse was defined as follows: for a participant with a pre-vaccination titer <1:8, the post-vaccination titer must be >=1:16, and for a participant with a pre-vaccination titer >=1:8, the post-vaccination titer must be at least 4-fold greater than the pre-vaccination titer. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 1 (pre-vaccination) and Day 31 (30 days post-vaccination on Day 1)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 200 | 221
percentage of participants
  Serogroup A | 81.5 [75.4 to 86.6] | 66.5 [59.9 to 72.7]
  Serogroup C | 99.5 [97.2 to 100] | 97.7 [94.8 to 99.3]
  Serogroup Y | 96.5 [92.9 to 98.6] | 95.5 [91.8 to 97.8]
  Serogroup W | 94.5 [90.4 to 97.2] | 95.5 [91.8 to 97.8]

5. Primary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the case report form (CRF) in terms of diagnosis and onset window post-vaccination. Immediate events were recorded to capture medically relevant unsolicited systemic AEs (including those related to the study vaccine administered) which occurred within the first 30 minutes after vaccination.
Time Frame: Up to 30 minutes post-vaccination on Day 1
Population: The safety analysis set (SafAS) included participants who received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 223 | 223
Participants | 0 | 1

6. Primary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. An injection site reaction was an AR at and around the injection site considered to be related to the study vaccine administered and were commonly inflammatory reactions. Systemic ARs were all ARs that were not injection site reactions and included systemic manifestations such as headache, fever, as well as localized or topical manifestations.
Time Frame: From the study vaccine administration (Day 1) up to 7 days post-vaccination, up to Day 8
Population: The SafAS included participants who received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 223 | 223
Participants
  Solicited injection site reactions | 29 | 29
  Solicited systemic reactions | 34 | 24

7. Primary Outcome: Number of Participants With Unsolicited Non-Serious Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: From the study vaccine administration (Day 1) up to 30 days post-vaccination (Day 31)
Population: The SafAS included participants who received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 223 | 223
Participants | 48 | 11

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An SAE was any AE that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was other medically important event. An AESI (serious or non-serious) was one of scientific and medical concern specific to the Sponsor's study vaccine or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor was appropriate.
Time Frame: From the study vaccine administration (Day 1) up to 30 days post-vaccination (Day 31)
Population: The SafAS included participants who received the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
Number analyzed (Participants) | 223 | 223
Participants
  SAEs | 3 | 2
  AESIs | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs, SAEs and all-cause mortality (deaths) were collected from the study vaccine administration (Day 1) up to 30 days post-vaccination (Day 31)
Description: Analysis was performed on the SafAS.
Arm/Group | MenACYW Conjugate Vaccine: 12-23 Months of Age | MenACYW Conjugate Vaccine: 24 Months of Age and Above
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/223
Serious Adverse Events (participants affected / at risk) | 3/223 | 2/223
Other Adverse Events (participants affected / at risk) | 59/223 | 39/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW Conjugate Vaccine: 12-23 Months of Age (N=223) | MenACYW Conjugate Vaccine: 24 Months of Age and Above (N=223)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW Conjugate Vaccine: 12-23 Months of Age (N=223) | MenACYW Conjugate Vaccine: 24 Months of Age and Above (N=223)
Upper Respiratory Tract Infection (Infections and infestations) | 22 (22) | 2 (2)
Injection Site Erythema (General disorders) | 13 (13) | 11 (11)
Injection Site Pain (General disorders) | 26 (26) | 23 (23)
Pyrexia (General disorders) | 16 (16) | 7 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 17 (17) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 15 (15)
Crying (General disorders) | 13 (13) | 0 (0)
Malaise (General disorders) | 0 (0) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT06228586/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06228586/SAP_001.pdf